CLINICAL TRIAL: NCT07000981
Title: Predicting Fall Risk With Machine Learning and Computer Vision: Development of A Clinical Decision Support System in Nursing Care
Brief Title: AI-Powered Fall Risk Prediction in Nursing Care
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Ceviz, ACeviz [Ahmet CEVİZ] Principal Investigator, Inonu University
Other Study IDs: INONU-FN-AC-01
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Accidental Falls; Risk Assessment; Nursing Assessment; Machine Learning; Computer Vision

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to develop a nursing clinical decision support system for fall risk prediction using machine learning and computer vision techniques. The system is intended to offer advantages over traditional scales, including real-time analysis, contactless monitoring, objective evaluation, and personalized risk prediction-ultimately aiming to improve patient safety and reduce complications related to falls in clinical settings.

This study aims to answer the following questions:

Can machine learning models serve as valid tools for fall risk prediction?

Is the proposed system feasible for use in clinical environments?

Inclusion criteria for participants:

* Aged 18 years or older
* Able to read and write in Turkish
* Able to walk with or without assistance
* Willing to voluntarily participate in the study

Exclusion criteria:

* Inability to speak or understand Turkish adequately
* Being intubated
* Being physically restrained
* Being immobile
* Having a diagnosed cognitive impairment

Participants' basic information-including age, height, and weight-will be collected through a demographic data form. Fall risk will be initially assessed using the Morse Fall Scale. Then, a walking assessment will be conducted using a digital camera-based computer vision system as participants walk at a comfortable pace in a clinical corridor. Additionally, an accelerometer placed in the participants' pockets will record three-axis acceleration (X, Y, Z) during walking.

The data obtained will be analyzed using machine learning algorithms to estimate lower and upper limb biomechanics in real time. Features such as step length, cadence, gait cycle, and range of motion (ROM) will be extracted. These features, combined with Morse Fall Scale scores, will be used to train and validate an artificial neural network (ANN).

The study aims to contribute to the development of a reliable, objective, and real-time system capable of predicting fall risk in clinical environments through gait analysis.

DETAILED DESCRIPTION:
Type of Research:

This research is planned as Design and Development Research as an innovative system will be developed.

Place and Time of the Research:

The research will be conducted at the Physical Medicine and Rehabilitation department of a research hospital located in eastern Turkey between June and August 2025.

Population and Sample of the Study:

The study population consisted of all patients treated at the Physical Medicine and Rehabilitation Service at Turgut Özal Medical Center. The sample size for the study was determined to be 161 using a power analysis, with a confidence interval of 0.95, a bias level of 0.05, an effect size of 0.30, and a representativeness of 0.95.

Individuals who meet the inclusion criteria will be included in the sample of the study until the sample size is reached by non-probability sampling method.

General Framework:

The development of the fall risk assessment application in this study will follow a structured methodology. It begins with the selection of participants who meet the defined inclusion and exclusion criteria. For each participant, a descriptive information form will be created, including basic data such as age, height, weight, and other relevant variables. This information will be evaluated in conjunction with the Morse Fall Scale, which will be used to assess each participant's risk of falling. Patients included in the sample will first be assessed using the Morse Fall Scale, followed by a gait analysis. This gait assessment will be conducted using a computer vision system that employs a digital camera to monitor participants as they walk at a comfortable pace in a clinical corridor. Additionally, participants will carry an accelerometer in their pockets to record acceleration data along the X, Y, and Z axes during walking. The collected data will be processed in real time using machine learning techniques to estimate the biomechanics of the lower and upper limbs. Key gait features-such as stride length, cadence, gait period, and range of motion (ROM)-will be extracted. These features, along with Morse Fall Scale scores, will be used to train and validate an artificial neural network (ANN) designed to identify potential correlations between gait characteristics and fall risk levels.

As a result, the final system will be able to predict the fall risk of new cases in real time through gait analysis.

Computer Vision System:

The computer vision system will consist of one camera connected to a computer and will be configured to record at 20 frames per second (FPS). The camera will be mounted on a tripod to ensure stable imaging of all extremities. The system will be complemented by artificial illumination from infrared reflectors with a wavelength of 850 nm to ensure uniform illumination of the study area without disturbing the participants.

Walk Evaluation Protocol:

A biomechanical gait study will be performed using computer vision to determine kinematic parameters. The methodology used to obtain this information requires participants to move through the clinic corridor at their own comfort pace. Patients will also be able to walk with the help of a companion or nurse. They will be informed about this process in advance to ensure that it does not pose any risk to their health or safety. Each test can be interrupted at any time if the participant feels they need assistance due to fatigue, discomfort or dizziness

Biomechanics Prediction:

For image analysis, we will use You Only Look Once, version 8 (YOLOv8) , a high-speed, high-precision model used in computer vision. YOLOv8 supports tasks such as detection, segmentation, pose estimation, tracking and classification. This model can be trained using specialized databases to recognize specific objects such as humans and track key points. The development will be based on the placement of key points to indicate different segments of the left and right extremities. For the development of the algorithm, we have chosen to use the open-source Keras library in Python, designed for the training and implementation of deep learning models. These models can be used both for the development of neural networks for the analysis of statistical databases and for the training of models for the analysis of images performing tasks such as the detection of objects, people, faces and body orientation. Therefore, using the database obtained from Keras, the training of personalized models will be carried out, where information and images are divided for training and validation. The resulting model will then be used for the analysis of gait test videos. Here, each frame will be taken to perform the identification of each limb segment through key points

Machine Learning Based Classifiers:

In this study, four classifiers will be used to classify gait data, including convolutional neural network (CNN), long short-term memory (LSTM) neural network, support vector machine (SVM) and K-nearest neighbor (KNN) classifier. A CNN with two 2D convolutional layers will be used as a reference. CNN is a type of deep neural network classifier used in image classification and recognition. It can recognize features directly from the data instead of extracting them manually. In the CNN structure in this study, the data will be passed through various layers with different tasks. The input will be transferred to the convolution layer where a spatial filter is applied to the inputs in the form of a weight window. This approach has been used in medical applications where the datasets are small in size and has shown success in medical image recognition.

Data Collection:

The data will be collected in the Physical Medicine and Rehabilitation department of a research hospital located in eastern Turkey between June and August 2025. Data will be gathered by the researcher through questionnaires and measurements using the face-to-face interview method.

Data Collection Tools: Descriptive Information Form, Morse Fall Risk Scale, a camera with video capture feature and an accelerometer will be used to collect the data.

Descriptive Information Form: This form was prepared within the scope of the master's thesis titled "Computer Vision in Fall Risk Prediction with Machine Learning: Development of a Nursing Clinical Decision Support System". The aim of our study is to predict the fall risk of patients hospitalized in the neurology clinic with machine learning and computer vision methods.

Morse Falls Scale: Developed in 1985 by Janice M. Morse in a randomized controlled study with 100 falling patients and 100 non-falling patients, the Morse Falls Scale was adapted to Turkish by Demir and Intepeler in 2012. It is an effective and simple measurement tool that is frequently used in hospitals in Turkey and used to diagnose potential patient fall risks for the nursing profession. The scale consists of six criteria (secondary diagnosis, presence of a history of falls, mobilization support, presence of intravenous access or heparin use, gait/transfer, and mental status) that diagnose fall risk. According to this assessment tool, if the patient has a score below 25 points, he/she is in the low risk group for falls. If the score is between 25 and 50, the patient is in the medium risk group, and if the score is 51 and above, the patient is in the high risk group. A minimum score of 0 and a maximum score of 125 can be obtained from the scale. This scale allows a systematic determination of the fall risk of patients in clinical settings. While 82.9% of the nurses stated that the Morse Falls Scale was easy and quick to use, 54% of the nurses stated that they diagnosed potential fall risks by allocating less than three minutes to the patient while using this scale. Although the Cronbach's Alpha value of the original scale was 0.16, the Cronbach's Alpha value in the Turkish validity and reliability study was calculated as 0.55.

Video Recording: The spontaneous gait of the patients will be recorded for 2 minutes with a video recording device to create a database for computer vision and machine learning methods.

Accelerometer: This simple device is sized enough for patients to carry in their pockets and measures the accelerations of movement in the X, Y and Z axes during spontaneous walking. These measurements will be recorded and collected simultaneously with video recording for 2 minutes and will provide a database for the system to be created with the deep learning method.

Data Evaluation:

In this research, One-way Analysis of Variance (one-way ANOVA) with Post-hoc Least Significant Difference (PostHoc LSD) will be used to determine the statistical difference in the average range of motion of a joint between different gait patterns and the average gait pattern recognition accuracy between machine learning algorithms. Pearson chi-square or Bonferroni correction test will be performed to determine the difference in each gait shape recognition accuracy between multiple machine learning algorithms for different gait shapes. RStudio software will be used for statistical analysis. p value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Accepting voluntary participation in the study
* Be able to read and write Turkish
* Being able to walk with or without support

Exclusion Criteria:

* Not being able to speak or understand Turkish adequately
* Being intubated.
* To be identified.
* Being immobile
* Having a mental disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is planned to be conducted on patients who meet the inclusion criteria and are hospitalized in the Physical Medicine and Rehabilitation department of a research hospital located in the eastern region of Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Özden, Assistant Professor, Study Director — Inonu University
Locations (1):
- Turgut Özal Medical Center, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive health information, and there are no current plans or resources in place to support secure de-identification and controlled data access. Furthermore, the study protocol does not include provisions for data sharing.

REFERENCES:
- [Background] Akhtaruzzaman M, Shafie AA, Khan MR. Gait Analysis: Systems, Technologies and Significance. J Mech Med Biol. 2016;16(7).
- [Background] Demir NY, Intepeler ŞS. Adaptation Of Morse Fall Scale To Turkish And Determination Of Sensitivity And Specificity. J Ege Univ Nurs Fac. 2012;28(1):57-71.
- [Background] Zhao M, Chang CH, Xie W, Xie Z, Hu J. Cloud Shape Classification System Based on Multichannel CNN and Enhanced FDM. IEEE Access. 2020;8:44111-24.
- [Background] Krizhevsky A, Sutskever I, Hinton GE. ImageNet classification with deep convolutional neural networks. Commun ACM. 2017;60(6):84-90.
- [Background] Santos GL, Endo PT, Monteiro KHC, Rocha EDS, Silva I, Lynn T. Accelerometer-Based Human Fall Detection Using Convolutional Neural Networks. Sensors (Basel). 2019 Apr 6;19(7):1644. doi: 10.3390/s19071644. PMID 30959877
- [Background] Yunas SU, Ozanyan KB. Gait Activity Classification Using Multi-Modality Sensor Fusion: A Deep Learning Approach. IEEE Sens J. 2021;21(15):16870-9.
- [Background] Manssor SAF, Sun S, Elhassan MAM. Real-Time Human Recognition at Night via Integrated Face and Gait Recognition Technologies. Sensors (Basel). 2021 Jun 24;21(13):4323. doi: 10.3390/s21134323. PMID 34202659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included patients treated at the Department of Physical Medicine and Rehabilitation at Turgut Özal Medical Center. A priori power analysis indicated that a sample size of 161 participants would be sufficient to detect an effect size of 0.30 with 95% confidence and 5% margin of error. In total, 177 participants were enrolled using non-probability sampling to accommodate potential data loss during the study.
Pre-assignment Details: Research Inclusion Criteria
  * Being 18 years or older
  * Being able to read and write Turkish
  * Being able to walk with or without support Study Exclusion Criteria
  * Not being able to speak or understand Turkish at a sufficient level
  * Being diagnosed
  * Being immobile
  * Being cognitively inadequate for the study
Groups:
- Cohort Group: All 177 participants completed the fall risk assessment using the Decision Support System.
Period: Overall Study
Arm/Group | Cohort Group
Started | 177
Completed | 177
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort Group: The fall risk assessment application used in this study was developed using a methodology. A descriptive information form was created for each participant, including basic information such as age, height, weight, and other data. This information was then integrated into the Morse Fall Scale to assess fall risk. Patients included in the sample were first administered the Morse Fall Scale and then given a gait assessment using a computer vision system consisting of a digital camera that monitored patients walking at a comfortable pace in the clinic corridor. Acceleration along the X, Y, and Z axes during walking was also assessed using an accelerometer carried in the patients' pockets.
  Data obtained from this system was analyzed using machine learning methods to estimate the biomechanics of the lower and upper extremities in real time. Inferences were then drawn regarding key gait characteristics such as stride length, cadence, period, and range of motion. This data was then used to train and validate an artificial neural network (ANN) that sought correlations between the extracted features and the Morse Fall Scale score. As a result, the final system was able to predict the fall risk of new cases in real time through gait analysis. The AI-based system developed as part of the study was introduced to the literature under the name "GuArDrop."
Arm/Group | Cohort Group
Number analyzed (Participants) | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.38 (16.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 177
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.21 (5.64)

OUTCOME MEASURES:

1. Primary Outcome: Fall Risk Categories Based on the Morse Fall Scale
Description: Assessment of the patient's fall risk with the Morse Fall Scale It is an effective and simple measurement tool that is frequently used in hospitals in Turkey and used to diagnose potential patient fall risks for the nursing profession. The scale consists of six criteria (secondary diagnosis, presence of a history of falls, mobilization support, presence of intravenous access or heparin use, gait/transfer, and mental status) that diagnose fall risk. According to this assessment tool, if the patient has a score below 25 points, he/she is in the low risk group for falls. If the score is between 25 and 50, the patient is in the medium risk group, and if the score is 51 and above, the patient is in the high risk group. A minimum score of 0 and a maximum score of 125 can be obtained from the scale. This scale allows a systematic determination of the fall risk of patients in clinical settings.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort Group
Number analyzed (Participants) | 177
Participants
  Low Risk (<25) | 131
  Medium Risk (25-50) | 41
  High Risk (≥51) | 5

2. Primary Outcome: Fall Risk Classification Accuracy of the Decision Support System
Description: Classification accuracy of the decision support system was evaluated based on the percentage of test units correctly classified. The scale ranges from 0% to 100%, where higher values indicate better performance. This metric reflects the proportion of correctly identified cases by the system during model evaluation.
Time Frame: Day 1
Population: A total of 177 participants were enrolled in the study, out of which 35 were assigned to the test group for evaluating the model's classification performance. This test group was not used in the training or validation phases.
Measure: Mean (Standard Error); unit: Percentage (%)
Arm/Group | Cohort Group
Number analyzed (Participants) | 35
Percentage (%) | 91.4 (2.10)

3. Primary Outcome: Classification Performance Metrics of the Decision Support System (F1 Score, Precision, Recall)
Description: This outcome measure evaluates the classification performance of a clinical decision support system using standard machine learning metrics: precision, recall, and F1-score. These metrics are based on a scale ranging from 0 to 1. Higher values indicate better classification performance. Precision is defined as the proportion of true positive predictions among all positive predictions. Recall is defined as the proportion of true positive predictions among all actual positives. The F1-score is the harmonic mean of precision and recall.
Time Frame: Day 1
Population: Of the 177 enrolled participants, 35 were allocated to the test group for the evaluation of model performance using standard machine learning metrics. The remaining participants were used for model training and validation.
Measure: Mean (Standard Error); unit: Proportion
Arm/Group | Cohort Group
Number analyzed (Participants) | 35
Proportion
  Precision (AUC) | 0.864 (2.58)
  Recall | 0.914 (2.10)
  F1-Score | 0.920 (2.03)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Cohort Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT07000981/Prot_SAP_000.pdf